CLINICAL TRIAL: NCT00269568
Title: A Multicenter, Randomized Comparison of Mifepristone and Misoprostol Administered Simultaneously Versus 24 Hours Apart for Abortion Through 63 Days
Brief Title: Mifepristone at Same Time Multicenter Study
Acronym: MAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pittirb0404133
Record Dates: First submitted 2005-09-12; First posted 2005-12-23 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Abortion Seekers
Keywords: medical abortion; mifepristone; misoprostol
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mifepristone and misoprostol

SUMMARY:
This is a multicenter, randomized study. 564 healthy women, age 18 years or older, with an intrauterine pregnancy, and requesting a medical abortion, will be recruited to participate in this prospective clinical trial. This study will provide an evaluation of oral mifepristone 200 mg and vaginal misoprostol 800 mcg administered simultaneously in women up to 63 days gestation. The aims of the study are to compare the complete abortion rates, at 7 and 14 days after misoprostol administration, when using mifepristone 200 mg orally and misoprostol 800 mcg vaginally are administered simultaneously and 24 hours apart in women up to 63 days gestation. Assessment of side effects (nausea, vomiting, pain) as well as acceptability will be done using pre and post-study questionnaires, and visual analogue scales. Complete abortion rate within 24 hours is expected to be 90%

DETAILED DESCRIPTION:
This is a multicenter, randomized study. 564 healthy women, age 18 years or older, with an intrauterine pregnancy, and requesting a medical abortion, will be recruited to participate in this prospective clinical trial. This study will provide an evaluation of oral mifepristone 200 mg and vaginal misoprostol 800 mcg administered simultaneously in women up to 63 days gestation. The aims of the study are to compare the complete abortion rates, at 7 and 14 days after misoprostol administration, when using mifepristone 200 mg orally and misoprostol 800 mcg vaginally are administered simultaneously and 24 hours apart in women up to 63 days gestation. Assessment of side effects (nausea, vomiting, pain) as well as acceptability will be done using pre and post-study questionnaires, and visual analogue scales. Complete abortion rate within 24 hours is expected to be 90%.

ELIGIBILITY:
Inclusion Criteria:pregnancy equal to or less than 63 days at enrollment -

Exclusion Criteria:abnormal pregnancy diagnosed by ultrasound

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1128 (Actual)
Dates: Start 2004-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
complete abortion rate | 5 weeks after treatment

SECONDARY OUTCOMES:
to compare complete abortion rates by gestational age | 5 weeks after treatment
compare bleeding and side effect profiles | up to 5 weeks after treatment
compare acceptability of the two regimens | 2 weeks after treatment
compare the expression of EP3 receptor mRNA in cervical tissue 2 and 24 hours after mifepristone treatment to pretreatment control | up to 24 hours after treatment
measure time to first ovulation | up to 10 weeks after treatment
compare elapsed time to ovulation between treatment regimens | up to 10 weeks after treatment
evaluate continuation rates of combined hormonal contraceptives in women with immediate initiation versus traditional Sunday start | up to 12 weeks after treatment
describe the prevalence of domestic violence in a medical abortion research population | at time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Creinin, MD, Principal Investigator — Universtity of Pittsburgh
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Oregon Health Sciences University, Portland, Oregon
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Creinin MD, Schreiber CA, Bednarek P, Lintu H, Wagner MS, Meyn LA; Medical Abortion at the Same Time (MAST) Study Trial Group. Mifepristone and misoprostol administered simultaneously versus 24 hours apart for abortion: a randomized controlled trial. Obstet Gynecol. 2007 Apr;109(4):885-94. doi: 10.1097/01.AOG.0000258298.35143.d2. PMID 17400850
- [Result] Bednarek PH, Nichols MD, Carlson N, Edelman AB, Creinin MD, Truitt S, Jensen JT. Effect of "observed start" vs. traditional "Sunday start" on hormonal contraceptive continuation rates after medical abortion. Contraception. 2008 Jul;78(1):26-30. doi: 10.1016/j.contraception.2008.02.012. Epub 2008 May 6. PMID 18555814